CLINICAL TRIAL: NCT00940576
Title: Dietetic Effects of Mare's Milk in Patients With Chronic Inflammatory Bowel Diseases (IBD) - a Double Blind Placebo Controlled Cross-over Study.
Brief Title: Dietetic Efficacy of Mare's Milk for Patients With Chronic Inflammatory Bowel Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Gerhard Jahreis, Prof. Dr., University of Jena
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LSEP_H08b-00
Record Dates: First submitted 2009-07-15; First posted 2009-07-16 (Estimated); Results first posted 2015-04-20 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Ulcerative Colitis; Crohns Disease
Keywords: mare's milk, Crohn's disease, ulcerative colitis, clinical
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mare´s milk (Experimental): oral intake of of 250 ml mare´s milk
  Interventions: Dietary Supplement: mare´s milk; Other: placebo drink
- placebo drink (Placebo Comparator): oral intake of of 250 ml placebo drink
  Interventions: Dietary Supplement: mare´s milk; Other: placebo drink

INTERVENTIONS:
Dietary Supplement: mare´s milk — oral intake of 250 ml mare's milk first, then placebo drink daily during 8 weeks of each (cross over design)
Other: placebo drink — oral intake of 250 ml placebo drink first, then mare's milk daily during 8 weeks of each (cross over design)

SUMMARY:
Mare's milk consumption could improve the well-being in patients with Crohn's disease and ulcerative colitis, respectively.

DETAILED DESCRIPTION:
Background: Dietetic effects of mare's milk have been reported for a long time and can be based on bactericidal and immunological components of mare's milk.

Objective: Dietetic effects of oral intake of mare's milk in adolescent patients with chronic inflammatory bowel diseases were investigated.

Design: In a randomized, placebo-controlled, double-blind, cross-over intervention study, eight Crohn's disease patients and nine ulcerative colitis patients received daily 250 mL mare's milk or placebo drink.

ELIGIBILITY:
Inclusion Criteria:

clear and definite diagnosis of ulcerative colitis and Crohn's disease resp.

Exclusion Criteria:

lactose intolerance and pregnancy

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2000-07; Primary Completion 2001-02 (Actual); Study Completion 2001-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Jahreis, Prof. Dr., Principal Investigator — Professor in Ordinary
Locations (2):
- Germany (2):
  - Friedrich Schiller University Jena, Department of Nutritional Physiology, Jena, Thuringia
  - University of Jena, Institute of Nutrition, Department of Nutritional Physiology, Jena, Thuringia

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Intake of Mare´s Milk First, Then Placebo: Oral Intake of 250 ml per day Mare´s Milk First, Then 250 ml per day Placebo
- Oral Intake of Placebo First, Then Mare´s Milk: Oral intake of 250 ml per day placebo first, then 250 ml per day mare´s milk
Period: Overall Study
Arm/Group | Oral Intake of Mare´s Milk First, Then Placebo | Oral Intake of Placebo First, Then Mare´s Milk
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Oral intake of placebo first, then mare´s milk and oral intake of mare´s milk first, then placebo respectively.
Arm/Group | All Study Participants
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.0 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 7
Region of Enrollment [Number; unit: participants]
  Germany | 17

OUTCOME MEASURES:

1. Secondary Outcome: Extra-intestinal Pain
Description: The patients recorded daily their extraintestinal disorders (fever, anal fissures, stomatitis, arthralgia, skin irritation) using a treatment improvement protocol (TIP).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Percentage of days with pain
Groups:
- Entire Study Population: oral intake of 250 ml mare´s milk or placebo drink daily
Arm/Group | Entire Study Population
Number analyzed (Participants) | 17
Percentage of days with pain
  Baseline | 28 (14)
  Start of placebo | 37 (25)
  End of placebo | 29 (15)
  Start of mare´s milk | 29 (15)
  End of mare´s milk | 10 (2)

2. Primary Outcome: Score of Crohn´s Disease and/or Ulcerative Colitis
Description: score for Crohn´s disease: Crohn´s Disease Activity Index (CDAI), < 150 = remission, 151-220 = moderate activity, 221-450 = severe activity; score for ulcerative colitis: Colitis Activity Index (CAI), 0-4 = remission, 5-9 = low activity, 10-16 = moderate activity, 17-23 = high activity.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients Crohn´s Disease | Patients Ulcerative Colitis
Number analyzed (Participants) | 8 | 9
units on a scale
  Baseline | 58 (20) | 1.8 (2.2)
  Start of placebo | 43 (16) | 1.2 (1.6)
  End of placebo | 51 (20) | 1.8 (2.3)
  Start of mare´s milk | 57 (22) | 1.7 (2.4)
  End of mare´s milk | 54 (16) | 2.8 (3.1)

ADVERSE EVENTS:
Time Frame: The period in which adverse event data were collected were 3 month.
Groups:
- Group 1: oral intake of 250 ml mare's milk daily
- Group 2: oral intake of 250 ml placebo daily
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No